CLINICAL TRIAL: NCT01259583
Title: Carbon Dioxide Insufflation (CO2) and Warm Water Infusion (WWI) Versus Standard Air Insufflation (AI) for Unsedated Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Arnaldo Amato, Doctor, Valduce Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CO2-01
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Warm Water; CO2 Colonoscopy; Unsedated Colonoscopy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- CO2 (Experimental): CO2 insufflation instead air insufflation in unsedated colonoscopy
  Interventions: Procedure: CO2
- Warm Water irrigation (Experimental): warm water irrigation during the insertion phase of colonoscopy
  Interventions: Procedure: Warm water

INTERVENTIONS:
Procedure: CO2 — CO2 insufflation
  Arms: CO2
Procedure: Warm water — warm water irrigation
  Arms: Warm Water irrigation

SUMMARY:
Due to the increasing demand for colonoscopy in clinical practice, great interest has recently renewed for unsedated colonoscopy. Both Carbon dioxide Insufflation (CO2) and Warm Water Infusion (WWI) have been advocated to improve patient tolerance for colonoscopy as compared to standard Air Insufflation (AI). This study is aimed at evaluating the performance of the above techniques versus AI in unsedated patients.

ELIGIBILITY:
Inclusion Criteria

* adult outpatients willing to undergo colonoscopy without routine initial sedation

Exclusion Criteria:

* refuse to initiate colonoscopy without routine sedation
* inadequate bowel preparation
* incapacity to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
number of patients undergoing complete unsedated colonoscopy | 6 months

SECONDARY OUTCOMES:
evaluation of pain and tolerability scores | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Valduce Hospital - Gastroenterology Department, Como, Italy

REFERENCES:
- [Derived] Amato A, Radaelli F, Paggi S, Baccarin A, Spinzi G, Terruzzi V. Carbon dioxide insufflation or warm-water infusion versus standard air insufflation for unsedated colonoscopy: a randomized controlled trial. Dis Colon Rectum. 2013 Apr;56(4):511-8. doi: 10.1097/DCR.0b013e318279addd. PMID 23478620